CLINICAL TRIAL: NCT00619632
Title: Boosting Breastfeeding in Low-Income, Multi-ethnic Women: A Primary Care Based RCT
Acronym: BINGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Montefiore Medical Center (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Karen Bonuck, PI, Albert Einstein College of Medicine
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 06-08-364; NIH R01 HD04976301A2; Montefiore IRB= 06-08-364
Record Dates: First submitted 2008-02-04; First posted 2008-02-21 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Breastfeeding; Breastfeeding, Exclusive
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): LC- Primary-care based lactation consultant meeting women pre- and post-natally.
  Interventions: Behavioral: Lactation Consultant
- 2 (Experimental): Provider Prompt
  Interventions: Behavioral: Provider Prompt
- 3 (Experimental): LC+Provider Prompt
  Interventions: Behavioral: LC+ Provider Prompt
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Lactation Consultant — Lactation consultant- primary care based, meets with women pre-natally, in the hospital, and at home up to 6 months post-partum.
  Arms: 1
Behavioral: Provider Prompt — Prompt in electronic prenatal record will appear 5 times throughout pregnancy re: up to 10 open-ended discussion points for provider to raise
  Arms: 2
Behavioral: LC+ Provider Prompt — Participants in this group receive both the LC and Provider Prompt interventions.
  Arms: 3

SUMMARY:
This is a randomized, controlled, single-center, single-blind, 2x2 factorial design trial of routine provider, primary care-based interventions to increase breastfeeding intensity up to 6 months in low-income multiethnic women, with stratification for maternal country of birth. The Best Infant Nutrition for Good Outcomes (BINGO) trial will randomize women into one of four treatment groups: (a) Prenatal Care Provider (PNC); (b) Lactation Consultant (LC); (c) PNC + LC, or; (d) Control. Thus, the separate and synergistic effects of the interventions will be tested, compared to a Control standard of care. The intervention and design build upon our prior trial of an LC intervention alone.

PNCs- certified nurse midwives and ob/gyns-- will use a brief, electronically prompted protocol with women in the PNC, and PNC + LC groups throughout pregnancy. An LC will arrange pre-natal one-on-one meetings, daily hospital, and home visits with women in the LC and PNC+LC groups. Descriptive data on infant health visits, and participant/provider experiences will be collected as secondary outcomes. Interviews at 1,3 and 6 months post-partum will collect infant feeding, and health visit data outside the medical center. Medical center visit data will be obtained from MIS data.

Primary Outcomes (Hypotheses): Breastfeeding

1. Breastfeeding Intensity at 1,3, and 6 Months
2. Exclusive Breastfeeding at 1,3, and 6 Months

   Secondary Outcomes (Descriptive): Infant Health, and Participant/Provider Experience
3. To describe the frequency and timing of infant health visits for "breast-feeding sensitive" illnesses
4. To describe participant and provider (LC and PNC) experience of the interventions.

DETAILED DESCRIPTION:
Primary Outcomes (Hypotheses): Breastfeeding

1. Breastfeeding Intensity at 1,3, and 6 Months- There will be significant differences in breastfeeding intensity among the 4 treatment groups. We expect that intensity will be greatest in the PNC+LC group, followed by the LC, then the PNC, and Control groups, respectively. Intensity will be assessed via 7 day recall of the frequency of breastmilk feedings vs. other liquids and solids.
2. Exclusive Breastfeeding at 1,3, and 6 Months- There will be significant differences in the rate of exclusive breastfeeding among the 4 treatment groups. We expect that rates of exclusive breastfeeding will be greatest in the PNC+LC group, followed by the LC, then the PNC, and Control groups, respectively.

   Secondary Outcomes (Descriptive): Infant Health, and Participant/Provider Experience
3. To describe the frequency and timing of infant health visits for "breast-feeding sensitive" illnesses (i.e., otitis media, gastrointestinal, and respiratory infections) by treatment group.
4. To describe the frequency and timing of infant health visits for "breast-feeding sensitive" illnesses by intensity of breastfeeding regardless of group assignment.
5. To describe participant and provider (LC and PNC) experience of the interventions.

BINGO is the first RCT in the US of routine provider, primary-care based interventions to increase breastfeeding (BF). Government task forces in the US3 and Canada specifically call for such trials, as well as trials to assess independent effects of combined interventions. BINGO is the first trial to apply strategies derived from the current National Breastfeeding Awareness Campaign (NBAC). BINGO will employ the NBAC message-- that exclusive BF for 6 months reduces infant ear infections, diarrhea, respiratory illness, and perhaps childhood obesity. We expect this message will yield greater BF intensity, and thus progress toward pending Healthy People 2010 goals for exclusive BF.

BINGO uses evidence-based strategies in practice, consistent with the NIH roadmap. Its interventions are logistically and economically sustainable in clinical practice. They support women pre- and post-natally, across multiple care settings (clinic, hospital, home). Both Certified Nurse Midwives and Ob/Gyns, deliver the PNC intervention, thus increasing generalizability. BINGO now has the enthusiastic support of perinatal nursing, physician, and lactation specialist groups. This support, at the outset, provides the foundation for effective BINGO interventions to be translated into practice.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled/plan to remain in care at the site throughout their pregnancy
* 1st or 2nd trimester (randomization will include trimester as a blocking factor)
* Aged 18 or older
* Can provide a reliable phone number and at least 2 alternative contacts
* Are carrying a singleton pregnancy
* Can communicate in English or Spanish

Exclusion Criteria:

* High risk of prematurity/NICU (e.g., ESRD, multiple prior preterms, congenital anomalies)
* Medical/obstetrical complications for which BF is or may be perceived to be contra-indicated (e.g., HIV+, HTLV-1, breast reduction surgery, Hepatitis B and C, pre-gestational diabetes )
* On chronic medications incompatible with BF (e.g., hypoglycemics, lithium, ciprofloxacin)
* Enrolled in site's Group Pre-natal Care (app. 60 women/year)
* Previously enrolled in MILK study
* Craniofacial or neurological conditions that prevent an infant from BF (post-partum exclusion)
* Reported use of street drugs (responds to reviewer comment of how to control for this)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 666 (Actual)
Dates: Start 2008-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Breastfeeding duration and intensity | Assessed at 1,3, and 6 months

SECONDARY OUTCOMES:
Infant health visits | 12 months
Patient and provider experiences of the interventions | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen A. Bonuck, PhD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Comprehensive Family Care Center, The Bronx, New York, United States

REFERENCES:
- [Derived] Bonuck K, Stuebe A, Barnett J, Labbok MH, Fletcher J, Bernstein PS. Effect of primary care intervention on breastfeeding duration and intensity. Am J Public Health. 2014 Feb;104 Suppl 1(Suppl 1):S119-27. doi: 10.2105/AJPH.2013.301360. Epub 2013 Dec 19. PMID 24354834
- [Derived] Andaya E, Bonuck K, Barnett J, Lischewski-Goel J. Perceptions of primary care-based breastfeeding promotion interventions: qualitative analysis of randomized controlled trial participant interviews. Breastfeed Med. 2012 Dec;7(6):417-22. doi: 10.1089/bfm.2011.0151. Epub 2012 May 23. PMID 22621223